CLINICAL TRIAL: NCT02453802
Title: Comparison of Topical and Infusion Tranexamic Acid on Blood Loss and Risk of Deep Vein Thrombosis After Total Knee Arthroplasty
Brief Title: Comparison of Topical and Infusion Tranexamic Acid After Total Knee Arthroplasty
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Wang Jun-Wen, Clinical Professor, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CMRPG8D1051
Record Dates: First submitted 2015-05-04; First posted 2015-05-27 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Osteoarthritis, Knee
Keywords: Tranexamic Acid; Total Knee Arthroplasty; Rivaroxaban
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Tranexamic Acid; Tranylcypromine; Rivaroxaban; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Topic TXA group (Active Comparator): Primary total knee replacement with intravenous 0.9% normal saline (20 ml) administration before deflation of the tourniquet and intraarticular application of Tranexamic Acid 5%,5ml/amp 3g (60ml) in 100 ml normal saline into knee joint after closure of the joint capsule
  Oral rivaroxaban (10mg) QD on PostOp Day 1 to 14 for VTE prophylaxis
  Interventions: Drug: Tranexamic Acid 5%,5ml/amp; Drug: rivaroxaban (10mg); Drug: 0.9% Normal Saline
- IV TXA group (Active Comparator): Primary total knee replacement with 1 g Tranexamic Acid 5%,5ml/amp administrated intravenously before deflection of the tourniquet and topical 160 ml 0.9% normal saline application after closure of joint capsule.
  Oral rivaroxaban (10mg) QD on PostOp Day 1 to 14 for VTE prophylaxis
  Interventions: Drug: Tranexamic Acid 5%,5ml/amp; Drug: rivaroxaban (10mg); Drug: 0.9% Normal Saline
- Control group (Placebo Comparator): Primary total knee replacement with 0.9% normal saline administration intravenously before deflation of the tourniquet and topical 160 ml 0.9% normal saline application after closure of joint capsule.
  Oral rivaroxaban (10mg) QD on PostOp Day 1 to 14 for VTE prophylaxis
  Interventions: Drug: rivaroxaban (10mg); Drug: 0.9% Normal Saline

INTERVENTIONS:
Drug: Tranexamic Acid 5%,5ml/amp — Intraarticular application of tranexamic acid 3g (60ml) in 100 ml normal saline into knee joint after closure of the joint capsule
  Other Names: Transamine
  Arms: Topic TXA group
Drug: Tranexamic Acid 5%,5ml/amp — IV TXA group: Primary total knee replacement with 1 g tranexamic acid administrated intravenously before deflection of the tourniquet
  Other Names: Transamine
  Arms: IV TXA group
Drug: rivaroxaban (10mg) — Oral rivaroxabam (10mg) QD on PostOp Day 1 to 14.
  Other Names: Xarelto
Drug: 0.9% Normal Saline — Primary total knee replacement with intravenous normal saline (20 ml) administration before deflation of the tourniquet
  Other Names: 0.9% sodium chloride
  Arms: Control group; Topic TXA group
Drug: 0.9% Normal Saline — Topical 160 ml normal saline application after closure of joint capsule.
  Other Names: 0.9% sodium chloride
  Arms: Control group; IV TXA group

SUMMARY:
The purpose of the study, therefore, is to conduct a prospective randomized controlled trial to investigate the blood-conservation effect of TXA in different TKA patients groups with rivaroxaban for VTE prophylaxis, first group by topical application, second group by infusion and a third group of placebo and observe whether there is difference in the occurrence of venous thromboembolism in those patient groups by venographic study

DETAILED DESCRIPTION:
Investigators previous experiences in minimally invasive (MIS) TKA showed that intraoperative infusion of TXA reduced 45% of postoperative blood loss and needs for transfusion from 20% to 4%. However, most of the orthopedic surgeons still hesitate to use TXA systemically in TKAs especially in high risk patients with a potential increase in thromboembolic events following surgery.

Because of this concern, recently, there were few reports demonstrating the cost-effectiveness of topical application of TXA in TKA patients. However, most of the reports compared the topical TXA with placebo in TKA patients, not with intravenous TXA. Recently, Georgiadis et al. conducted a double-blind, randomized controlled clinical trial are demonstrated similar transfusion rate and perioperative blood loss between topical administration and intravenous injection of TXA in TKA patients. There were no significant safety differences between the two groups. Low-molecular weight heparin (LMWH) was used for thromboembolism prophylaxis in that study.

Recently, chemical VTE prophylaxis such as rivaroxaban has been approved as a standard care after TKA because of its superior convenience and efficacy on VTE prophylaxis to LMWH in TKAs. However, because of direct blockage of the formation of thrombin from prothrombin by rivaroxaban, an increased postoperative bleeding has been reported. There have been little studies investigating the blood-conservation effect of TXA on TKA patients either by infusion or by topical application when rivaroxaban used as VTE prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

* End-stage arthritis of the knee
* Failure of medical treatment or rehabilitation
* Hemoglobin > 10g/dl
* No use of non-steroid anti-inflammatory agent one week before operation

Exclusion Criteria:

* Preoperative Hemoglobin ≦10 g/dl
* History of infection or intraarticular fracture of the affective knee
* Renal function deficiency (GFR < 55 ml/min/1.73m2)which is relative contraindicated for venography
* Elevated liver enzyme, history of liver cirrhosis, impaired liver function and coagulopathy (including long-term use anticoagulant)
* History of deep vein thrombosis, ischemic heart disease or stroke

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-05 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of any deep-vein thrombosis, non-fatal pulmonary embolism, or all-cause mortality | within 15 days after surgery (2 days after the last dose of rivaroxaban )
  Primary efficacy outcome is the composite of any deep-vein thrombosis, non-fatal pulmonary embolism, or all-cause mortality
Incidence of major bleeding after the first dose of rivaroxaban and all death related to postoperative bleedings | within 15 days after surgery (2 days after the last dose of rivaroxaban )
  Primary safety outcome is the composite of major bleeding after the first dose of rivaroxaban and all death related to postoperative bleedings Major bleeding was defined as bleeding that was fatal, that involved a critical organ, or that required reoperation or clinically overt bleeding outside the surgical site that was associated with a decrease in the hemoglobin level of 2 g or more per deciliter or requiring infusion of 2 or more units of blood

SECONDARY OUTCOMES:
Incidence of major venous thromboembolism | within 15 days after surgery (2 days after the last dose of rivaroxaban )
  the secondary efficacy outcomes include major venous thromboemolism defined as the composite of proximal deep-vein thrombosis, non-fatal pulmonary embolism, and VTE related death
Secondary safety outcome was composite of any non-major bleeding and all wound complications after operation | within 15 days after surgery (2 days after the last dose of rivaroxaban )
  non-major bleeding including hemorrhagic wound complications (excessive wound hematoma or bleeding at the surgical site
Incidence of wound complications after surgery | within 30 days of the procedure
  composite of hematoma, superficial wound infection, and deep infection requiring return to surgery
Total blood loss after surgery | From the operation to the postoperative day 4
  Total blood loss was calculated according to Nadler et al., which used maximum postoperative reduction of the Hb level adjust for weight and height of the patient. The formula is as follows, Total blood loss = (Total blood volume x [change in Hb level / preoperative Hb level])x1000+volume transfused.

OTHER OUTCOMES:
Incidence of venographic positive deep-vein thrombosis (any, proximal, distal) | on the second day after last dose of rivaroxaban (postoperative day 15)
Incidence of positive finding of pulmonary embolism by computed tomography | on the second day after last dose of rivaroxaban (postoperative day 15)

CONTACTS AND LOCATIONS:
Overall Officials: Jun-Wen Wang, MD, Study Chair — Chang Gung Memorial Hospital
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Koahsiung, Taiwan, Taiwan

REFERENCES:
- [Background] Gomez-Barrena E, Ortega-Andreu M, Padilla-Eguiluz NG, Perez-Chrzanowska H, Figueredo-Zalve R. Topical intra-articular compared with intravenous tranexamic acid to reduce blood loss in primary total knee replacement: a double-blind, randomized, controlled, noninferiority clinical trial. J Bone Joint Surg Am. 2014 Dec 3;96(23):1937-44. doi: 10.2106/JBJS.N.00060. PMID 25471907
- [Background] Lin PC, Hsu CH, Chen WS, Wang JW. Does tranexamic acid save blood in minimally invasive total knee arthroplasty? Clin Orthop Relat Res. 2011 Jul;469(7):1995-2002. doi: 10.1007/s11999-011-1789-y. Epub 2011 Feb 1. PMID 21286886
- [Background] Lin PC, Hsu CH, Huang CC, Chen WS, Wang JW. The blood-saving effect of tranexamic acid in minimally invasive total knee replacement: is an additional pre-operative injection effective? J Bone Joint Surg Br. 2012 Jul;94(7):932-6. doi: 10.1302/0301-620X.94B7.28386. PMID 22733948
- [Background] Wind TC, Barfield WR, Moskal JT. The effect of tranexamic acid on blood loss and transfusion rate in primary total knee arthroplasty. J Arthroplasty. 2013 Aug;28(7):1080-3. doi: 10.1016/j.arth.2012.11.016. Epub 2013 Mar 28. PMID 23541868
- [Background] Chimento GF, Huff T, Ochsner JL Jr, Meyer M, Brandner L, Babin S. An evaluation of the use of topical tranexamic acid in total knee arthroplasty. J Arthroplasty. 2013 Sep;28(8 Suppl):74-7. doi: 10.1016/j.arth.2013.06.037. PMID 24034510
- [Background] Konig G, Hamlin BR, Waters JH. Topical tranexamic acid reduces blood loss and transfusion rates in total hip and total knee arthroplasty. J Arthroplasty. 2013 Oct;28(9):1473-6. doi: 10.1016/j.arth.2013.06.011. Epub 2013 Jul 23. PMID 23886406
- [Background] Georgiadis AG, Muh SJ, Silverton CD, Weir RM, Laker MW. A prospective double-blind placebo controlled trial of topical tranexamic acid in total knee arthroplasty. J Arthroplasty. 2013 Sep;28(8 Suppl):78-82. doi: 10.1016/j.arth.2013.03.038. Epub 2013 Jul 29. PMID 23906869
- [Background] Lassen MR, Ageno W, Borris LC, Lieberman JR, Rosencher N, Bandel TJ, Misselwitz F, Turpie AG; RECORD3 Investigators. Rivaroxaban versus enoxaparin for thromboprophylaxis after total knee arthroplasty. N Engl J Med. 2008 Jun 26;358(26):2776-86. doi: 10.1056/NEJMoa076016. PMID 18579812
- [Background] Turpie AG, Lassen MR, Davidson BL, Bauer KA, Gent M, Kwong LM, Cushner FD, Lotke PA, Berkowitz SD, Bandel TJ, Benson A, Misselwitz F, Fisher WD; RECORD4 Investigators. Rivaroxaban versus enoxaparin for thromboprophylaxis after total knee arthroplasty (RECORD4): a randomised trial. Lancet. 2009 May 16;373(9676):1673-80. doi: 10.1016/S0140-6736(09)60734-0. Epub 2009 May 4. PMID 19411100
- [Background] Jameson SS, Rymaszewska M, Hui AC, James P, Serrano-Pedraza I, Muller SD. Wound complications following rivaroxaban administration: a multicenter comparison with low-molecular-weight heparins for thromboprophylaxis in lower limb arthroplasty. J Bone Joint Surg Am. 2012 Sep 5;94(17):1554-8. doi: 10.2106/JBJS.K.00521. PMID 22832942